CLINICAL TRIAL: NCT02695485
Title: Sensory Reconstruction in Different Region of the Digits: A Review of 151 Cases
Brief Title: Sensory Reconstruction of the Digits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Tangshan (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSZhao9012
Record Dates: First submitted 2016-02-19; First posted 2016-03-01 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Soft Tissue Defect of Digit
Keywords: dorsal digital island flap; sensory reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sensate flap (Other): the donor nerve harvested with the flap
  Interventions: Procedure: innervated sensate flap

INTERVENTIONS:
Procedure: innervated sensate flap — sensory reconstruction via digital nerve repair with the donor nerve of the flap

SUMMARY:
A retrospective study is conducted with 151 patients who has a soft tissue defect of digit treated with the sensate flaps from February 2005 to March 2014. Based on the different regions of soft tissue defects, the patients in the study are divided into four groups: (1) thumb group treated with the bilaterally innervated and traditional kite flaps; (2) distal finger group treated with the single- and dual-innervated dorsal digital flaps; (3) proximal finger group treated with heterodigital neurocutaneous island flap; and (4) awkward region group treated with Litter flap. The main outcomes are static 2-point discrimination and Semmes-Weinstein monofilament scores of the flap, and pain and patient satisfaction.

DETAILED DESCRIPTION:
At final follow-up, sensory restoration of the flap is measured using the static 2PD test and Semmes-Weinstein monofilament test. Using the visual analogue scale (VAS) that consists of a 10 cm line, patients are asked to report pain sensations of the recipient site. Patients report their satisfaction with functional recovery of the injured finger according to the Michigan Hand Outcomes Questionnaire that is based on a 5-point response scale.

ELIGIBILITY:
Inclusion Criteria:

* thumbtip degloving injury with a projecting tip of exposed bone or/and pulp defect; the defect ≥2 cm in length associated with the transected digital nerves in both sides; necessity to preserve thumb length; patient at or younger than 55 years of age

Exclusion Criteria:

* injury to the dorsum of the proximal or/and middle phalanx of the index finger; injury to the course of the FDMA; thumb nail bed defect; radial or ulnar portion of thumbtip or pulp defect

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 151 (Actual)
Dates: Start 2006-02; Primary Completion 2013-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Static 2PD test | 18 months to 24 months after surgery
  We use a Disk-Criminator to test two nearby points when touching the flap. It is often tested with two sharp points during a neurological examination and is assumed to reflect how finely innervated an area of flap is.
Pain sensation using the visual analogue scale | 18 months to 24 months after surgery
  Using the visual analogue scale (VAS) that consists of a 10 cm line, patients are asked to report pain sensations of the recipient site.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Chen C, Tang P, Zhang X. The dorsal homodigital island flap based on the dorsal branch of the digital artery: a review of 166 cases. Plast Reconstr Surg. 2014 Apr;133(4):519e-529e. doi: 10.1097/PRS.0000000000000016. PMID 24675204